CLINICAL TRIAL: NCT02484365
Title: The Accuracy of the Noninvasive Hemoglobin Monitoring for Preoperative Evaluation for Pediatric Patients
Brief Title: Preoperative Noninvasive Hemoglobin Monitoring in Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Yong-Hee Park, Assistant professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Other Study IDs: C2014202(1399)
Record Dates: First submitted 2015-03-06; First posted 2015-06-29 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Surgery
Keywords: Hemoglobins; Monitoring, Outpatient; Preoperative Period; Pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single arm study: No treatment or intervention will given to the patients
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — Attach adhesive probe on thumb or index finger

SUMMARY:
The preoperative evaluation including sampling blood in pediatric patients is hard to perform. However, the knowledge of the baseline cell blood count is important to prepare unexpected surgical bleeding etc.. The invasive procedure for blood sampling in small children is often failed and sometimes induces iatrogenic blood loss and parent's complaints. The Pulse Co-oximetry (Masimo) is recently developed device which can provide noninvasive hemoglobin value. However, the accuracy is controversial. There are studies in pediatric patients during surgery and in ICU. However, the comparison for preoperative evaluation is not analysed. Therefore, the investigators want to evaluate the accuracy for preoperative preparation in pediatric patients.

DETAILED DESCRIPTION:
There are not enough data comparing the noninvasive hemoglobin and venous hemoglobin in pediatric patients during preoperative period. The investigators will collect the venous sample and the noninvasive hemoglobin data from masimo within 1 hour. Without any additional medication, the patients will visit preanesthetic room and attach the probe of masimo on index finger. The R 20L or R25L will be used based on their weight. The parameter will be stabilized within 2 minutes and the SpHb and perfusion index will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1,2

Exclusion Criteria:

* Poor peripheral circulation
* Infection or trauma on the sensor contact region

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients age under 18 years planning to receive elective surgery under general anesthesia people live in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
hemoglobin | once, preoperative visit anesthetic office
  no F/U is needed

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Hee Park, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine : Chung-Aung University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jung YH, Lee J, Kim HS, Shin SH, Sohn JA, Kim EK, Choi JH. The efficacy of noninvasive hemoglobin measurement by pulse CO-oximetry in neonates. Pediatr Crit Care Med. 2013 Jan;14(1):70-3. doi: 10.1097/PCC.0b013e318260117d. PMID 23132397